CLINICAL TRIAL: NCT01473095
Title: A Phase 1 Dose Escalation Study of ARQ 092 in Adult Subjects With Advanced Solid Tumors and Recurrent Malignant Lymphoma
Brief Title: Phase 1 Dose Escalation Study of ARQ 092 in Adult Subjects With Advanced Solid Tumors and Recurrent Malignant Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 092-101
Record Dates: First submitted 2011-11-10; First posted 2011-11-17 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Solid Tumor; Malignant Lymphoma; Tumor
Keywords: AKT; ARQ 092; Targeted therapy; Molecular therapy; Biomarker; Phase 1; Phase I; Endometrial cancer; Lymphoma; AKT pathway; AKT signaling; AKT inhibitor; AKT pan inhibitor; AKT1; AKT2; AKT3; AKT1 mutation; AKT1-E17K; AKT1-E17K mutation; AKT 2 inhibitor; AKT 3 inhibitor; AKT 3 amplification; PI3K AKT mTOR signalling pathway; mTOR inhibitor; PI3K inhibitor; Clinical oncology; Tumor; Tumour; PIK3CA H1047R mutation
MeSH Terms: conditions — Lymphoma; Neoplasms; Endometrial Neoplasms | interventions — Miransertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ARQ 092 — Subjects in this study will receive ARQ 092 orally at dose levels specified for their respective dose cohorts. Dosing will begin at 10 mg every other day (QOD) and will escalate until the MTD or RP2D is determined. Cycles will be repeated in four-week (28 day) intervals until progression of disease, unacceptable toxicity, or another discontinuation criterion is met. In the case of toxicity, dose adjustment will be permitted.

SUMMARY:
This is an open-label, Phase 1, dose escalation study of oral ARQ 092 administered to subjects with advanced solid tumors and recurrent malignant lymphoma. The study is designed to explore the safety, tolerability, pharmacokinetics, and pharmacodynamics of ARQ 092 and to define a recommended Phase 2 dose of ARQ 092.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥18 years old
2. Histologically or cytologically documented, incurable, locally advanced or metastatic solid tumors or recurrent malignant lymphoma in subjects who failed standard therapy or for whom standard or curative therapy does not exist or is not tolerable.
3. Evaluable or measurable disease
4. Life expectancy greater than three months
5. ECOG performance status ≤2
6. Hemoglobin (Hgb) ≥9.5 g/dl
7. Absolute neutrophil count (ANC) ≥1.5 x 10^9/L
8. Platelet count ≥75 x 10^9/L
9. Total bilirubin ≤1.5 × upper limit of normal (ULN)
10. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3 × ULN
11. Serum creatinine ≤1.5 x ULN or creatinine clearance > 60 mL/min/1.73 m^2 for subjects with creatinine levels >1.5 x ULN
12. Agree to use double-barrier contraceptive measures or avoid intercourse during the study and for 90 days after the last dose of study drug

Exclusion Criteria:

1. History of Type 1 or 2 diabetes mellitus requiring regular medication (other than metformin or other oral hypoglycemic agents) or fasting glucose ≥160 mg/dL at the prestudy visit. If a diabetic cohort is enrolled, only subjects with a medical history of controlled Type 1 or 2 diabetes mellitus will be enrolled in the cohort.
2. Grade 2 or worse hypercholesterolemia or hypertriglyceridemia or >8% glycated Hb (HbA1C)
3. Malabsorption syndrome
4. Known brain metastases not radiographically stable for ≥3 months or leptomeningeal disease
5. History of myocardial infarction (MI) or NYHA Class II-IV congestive heart failure within 6 months of the administration of the first dose of ARQ 092 (MI occurring >6 months of the first dose of ARQ 092 will be permitted); Grade 2 or worse conduction defect (eg right or left bundle branch block); left ventricular ejection fraction (LVEF) < 50% assessed by echocardiogram/MUGA scan
6. Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within four weeks of the first dose of ARQ 092 (within 2 weeks for orally administered drugs)
7. Major surgery within four weeks of the first dose of ARQ 092
8. Previous treatment with AKT inhibitors
9. Concurrent severe uncontrolled illness not related to cancer
10. Ongoing or active known infection, including human immunodeficiency virus (HIV) infection or bleeding
11. Psychiatric illness/substance abuse/social situation that would limit compliance with study requirements.
12. Blood transfusion within 5 days prior to blood draw being used to confirm eligibility
13. Pregnant or breastfeeding
14. Previous other malignancy within 2 years prior to the first dose of ARQ 092, with the exception of carcinoma in-situ of the cervix, basal cell carcinoma and superficial bladder tumors curatively treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2017-07-06 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of ARQ 092 in subjects with advanced solid tumors and recurrent malignant lymphoma by monitoring frequency and severity of adverse events | Up to treatment discontinuation + 30 days with an estimated treatment duration of 4 to 16 weeks

SECONDARY OUTCOMES:
Assess the pharmacokinetic profile (Cmax, AUC, and half-life) of ARQ 092 | During the first 29 days of treatment for each dose level
Assess pharmacodynamic activity | During the first 29 days of treatment
Determine preliminary evidence of activity as defined by RECIST v 1.1 | Up to treatment discontinuation + 30 days with an estimated treatment duration of 4 to 16 weeks
Determine recommended Phase 2 dose | Up to treatment discontinuation + 30 days with an estimated treatment duration of 4 to 16 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Miami, Florida
  - Atlanta, Georgia
  - Lafayette, Indiana
  - San Antonio, Texas